CLINICAL TRIAL: NCT07277764
Title: Induction Therapy With High-Low Dose Radiotherapy Combined With Anti-PD-1 Monoclonal Antibody Followed by Definitive Radiotherapy in Recurrent Nasopharyngeal Carcinoma: A Single-Arm, Single-Center Phase II Trial
Brief Title: Induction High-Low Dose Radiotherapy Plus Anti-PD-1 Followed by Definitive Radiotherapy in Recurrent Nasopharyngeal Carcinoma (Single-Arm Phase II)
Acronym: REDEFINE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangxi Provincial Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REDEFINE
Record Dates: First submitted 2025-11-30; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Nasopharyngeal Carcinoma (NPC); Recurrent Nasopharyngeal Neoplasms
Keywords: recurrent NPC; re-irradiation; high-low dose radiotherapy; induction radio-immunotherapy; PD-1 inhibitor
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Nasopharyngeal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Induction High-Low Dose RT + Anti-PD-1 → Definitive RT → Anti-PD-1 Maintenance (Experimental): Induction: LD-RT 1.5 Gy ×3 (D1-D3) + HD boost 5 Gy ×3 to tumor core; Anti-PD-1 240 mg IV on D1 & D22. Definitive RT: from ~D28, IMRT 2 Gy ×28 (5 days/week) without concurrent IO. Maintenance: Anti-PD-1 240 mg IV Q3W up to 12 months. Early stop if CR at 50 Gy or ulcer occurs per protocol.
  Interventions: Radiation: High-Low Dose Radiotherapy

INTERVENTIONS:
Radiation: High-Low Dose Radiotherapy — Induction LD-RT 1.5 Gy ×3 (full lesion coverage) + HD boost 5 Gy ×3 (tumor core; carotid/mucosa sparing <3 Gy/fx); followed by definitive IMRT 2 Gy ×28.

SUMMARY:
This single-arm, single-center phase II trial evaluates the safety and efficacy of a non-continuous radio-immunotherapy strategy for recurrent nasopharyngeal carcinoma (NPC) unsuitable for surgery. Induction consists of three fractions of low-dose radiotherapy (1.5 Gy ×3) plus high-dose boosts (5 Gy ×3 to tumor core with carotid/mucosal sparing) combined with anti-PD-1 (240 mg IV on Day 1 and Day 22). After a 21-28-day interval, definitive IMRT (2 Gy ×28, 5 days/week) is delivered without concurrent immunotherapy to minimize immune damage. Anti-PD-1 maintenance (240 mg IV Q3W) starts within 2 weeks after radiotherapy for up to 12 months or until progression/toxicity. The primary endpoint is ORR at 3 months post-radiotherapy; secondary endpoints include 3-year OS, 3-year PFS, safety (NCI-CTCAE v5.0), and quality of life (EORTC QLQ-C30). Key eligibility: histologically confirmed non-keratinizing NPC (WHO II/III), rT2-rT4, ECOG 0-1, adequate organ function.

ELIGIBILITY:
Inclusion Criteria：

Histologically confirmed non-keratinizing NPC (WHO II/III); local (± regional) recurrence ≥1 year after prior radical therapy; surgery-ineligible;

rT2-rT4 (AJCC 8th); ECOG 0-1;

Adequate organ function (hematologic, hepatic, renal, coagulation per protocol thresholds);

Contraception requirements per protocol; signed informed consent.

Exclusion Criteria：

Distant metastasis at recurrence; active necrosis at recurrence; active/previous autoimmune disease; prior PD-1/PD-L1 therapy; uncontrolled comorbidities; active infections (HBV/HCV/HIV criteria per protocol); interstitial lung disease/pneumonitis; pregnancy/lactation; other protocol-specified exclusions.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2025-10-10 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR | 3 months after completion of definitive radiotherapy
  Objective Response Rate (ORR) at 3 months post-radiotherapy

SECONDARY OUTCOMES:
OS | 3 years.
  Overall Survival (OS) - Time from treatment start to death from any cause;
Progression-Free Survival | 3 years.
  Time from treatment start to progression or death;
Safety | through 12 months of therapy and 3-year follow-up.
  Incidence and grade of adverse events per NCI-CTCAE v5.0;

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangxi Cancer Hospital, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No